CLINICAL TRIAL: NCT05705752
Title: Effects on Balance of a Specific Training in Balance and Pilates: a Quasi-randomized Trial
Brief Title: Balance Training Vs Pilates Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández-Guillén, Assistant professor, PT, PhD, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BAL_VS_PIL
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Balance Training
Keywords: Pilates; Balance training; Physiotherapy; Prevention
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance (Experimental): Balance training group.
  Interventions: Other: Balance training
- Pilates (Active Comparator): Pilates group.
  Interventions: Other: Pilates training

INTERVENTIONS:
Other: Balance training — 12 sessions of balance training en 4 weeks, with a duration of 40-45 min each.
  Arms: Balance
Other: Pilates training — 12 sessions of Pilates training en 4 weeks, with a duration of 40-45 min each.
  Arms: Pilates

SUMMARY:
Many pathologies present balance disturbances, however, other types of therapies such as Pilates are increasingly used within the Physiotherapy profession. It is therefore necessary to know the effects that this type of exercise has compared to the traditional method of balance training in order to make good use of this type of therapy.

The objective of the study will be to know if there are differences between both types of training on the balance of the participants.

ELIGIBILITY:
Inclusion Criteria:

* University students between 18 and 35 years.

Exclusion Criteria:

* Diseases or patologies that affect balance.
* Professional sportmen.
* Having suffered an injury 6 months prior to the intervention.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Y Balance Test | 0 week
  The Y Balance Test (YBT) has the patient stand on one leg while reaching out in 3 different directions with the other lower extremity. They are anterior, posteromedial and posterolateral. When using the Y-Balance test kit, the 3 reaches yield a "composite reach distance" or composite score used to predict injury.
  The YBT showed good interrater test-retest reliability with an acceptable level of measurement error among multiple raters screening active duty service members, and a second study shows excellent reliability (ICC = 0.88- 0.99).
  An increase in the value of the test is indicative of the improvement of dynamic balance.
Y Balance Test | 5 week
  The Y Balance Test (YBT) has the patient stand on one leg while reaching out in 3 different directions with the other lower extremity. They are anterior, posteromedial and posterolateral. When using the Y-Balance test kit, the 3 reaches yield a "composite reach distance" or composite score used to predict injury.
  The YBT showed good interrater test-retest reliability with an acceptable level of measurement error among multiple raters screening active duty service members, and a second study shows excellent reliability (ICC = 0.88- 0.99).
  An increase in the value of the test is indicative of the improvement of dynamic balance.

SECONDARY OUTCOMES:
Emery test | 0 week, 5 week
  The single-leg Emery timed balance test was specifically designed to assess the balancing abilities of young people and adolescents. In this work, we conducted the eyes-closed dynamic test. The participants were asked to stand barefooted on an Airex® Balance-Pad with slight knee flexion of the weight-bearing limb and 45° degree flexion of the non-weight-bearing limb, keeping their hands on their hips. The timer was stopped when a participant lost their balance owing to one of the following situations: removal of hand from the hip; opening of the eyes; the non-weight-bearing limb touching the floor, the pad, or the weightbearing limb; or the pad or the foot of the non-weight-bearing limb moving from the initial test position. The longest duration of three attempts was recorded for each leg, allowing 30 s of rest between trials. Balance improves if time is increased on this test.

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández-Guillén, PT, PhD, Principal Investigator — University of Valencia
Locations (1):
- Faculty of Physiotherapy of the University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No